CLINICAL TRIAL: NCT00871780
Title: A Prospective, Open-label, Non-randomized, Clinical Trial to Determine if Natalizumab (Tysabri®) Improves Ambulatory Measures in Relapsing-remitting Multiple Sclerosis (RRMS) Patients "TIMER" Study
Brief Title: A Prospective, Open-label, Non-randomized, Clinical Trial to Determine if Natalizumab (Tysabri®) Improves Ambulatory Measures in Relapsing-remitting Multiple Sclerosis (RRMS) Patients
Acronym: TIMER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYS-IMA-08-11
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis (RRMS)
Keywords: TYSABRI naive; Relapsing-remitting multiple sclerosis (RRMS)
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab (Experimental): natalizumab 300 mg IV every 4 weeks for 48 weeks
  Interventions: Drug: BG00002 (natalizumab)

INTERVENTIONS:
Drug: BG00002 (natalizumab)
  Other Names: Tysabri®

SUMMARY:
The primary objective of the study is to evaluate the evolution of walking capacity as measured by the timed 100-meter walk test (T100T), timed 25-foot walk test (T25FW), maximum walking distance (MWD), and Expanded Disability Status Scale (EDSS) during the first year of therapy with natalizumab. The secondary objectives of this study are as follows:

* To evaluate the correlation between the MWD and EDSS and both walking tests, the T100T and the T25FW at Baseline, at Week 24 and at Week 48 of therapy.
* To determine how well each of the walking tests, T100T or T25FW, predicts walking limitations in all participants and in the subgroups of participants stratified by baseline EDSS.

ELIGIBILITY:
Key Inclusion Criteria:

* Must give written informed consent and provide all authorizations required by local law (for example, Protected Health Information [PHI])
* Men or women between 18 and 60 years of age, inclusive
* Must have Expanded Disability Status Scale (EDSS) less than or equal to 5.5 at baseline
* Must be able to walk at least 100 m without assistive devices
* Must be natalizumab-naïve
* Must have a documented diagnosis of a relapsing remitting form of multiple sclerosis (MS0 as defined by the revised McDonald Committee criteria (Polman et al., 2005)
* Must have had a recent (within 3 months from baseline) magnetic resonance imaging (MRI)
* Must have had at least 1 relapse in the previous year and must satisfy the locally approved therapeutic indications for Tysabri. If Tysabri is not yet approved in a specific country, patients must fulfill the following criteria:

  * Patients with high disease activity despite treatment with a beta-interferon defined as patients who have failed to respond to a full and adequate course of a beta-interferon
  * Patients must have had at least 1 relapse in the previous year while on therapy, and have at least 9 T2 hyperintense lesions in cranial MRI or at least 1 gadolinium (Gd)-enhancing lesion
  * Patients with rapidly evolving severe relapsing remitting multiple sclerosis defined as patients who have had 2 or more disabling relapses in one year and 1 or more Gd-enhancing lesions on brain MRI or significant increase in T2 lesions as compared to a previous MRI
* Must be stable in disability for at least 30 days prior to enrollment to the study
* Must be stable in symptomatic management of the disease, specifically spasticity, depression and fatigue for at least 30 days prior to enrollment to the study
* Must be considered by the Investigator to be free of signs and symptoms suggestive of progressive multifocal leukoencephalopathy (PML) based on medical history, physical examination, or laboratory testing
* Must be willing to discontinue and remain free from concomitant immunosuppressive or immunomodulatory treatment (including interferon [IFN] and glatiramer acetate [GA]) while being treated with natalizumab during the study.

Key Exclusion Criteria:

Unless otherwise specified, candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of the Screening Visit:

* Onset of a relapse within 50 days prior to first infusion
* Considered by the Investigator to be immunocompromised, based on medical history, physical examination, or laboratory testing or due to prior immunosuppressive treatment
* History of, or available abnormal laboratory results indicative of, any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric (including major depression), renal, and/or other major disease that would preclude the administration of a recombinant humanized antibody immunomodulating agent. The Investigator must re-review the subject's medical fitness for participation and consider any diseases that would preclude treatment
* History of malignancy (subjects with basal cell carcinoma that has been completely excised prior to study entry remain eligible)
* Known history of human immunodeficiency virus infection or hematological malignancy
* History of organ transplantation (including anti-rejection therapy)
* A clinically significant infectious illness (cellulitis, abscess, pneumonia, septicemia) within 30 days prior to the Screening Visit
* Treatment with immunosuppressant medications (mitoxantrone, cyclophosphamide, cyclosporine, azathioprine, methotrexate) within 6 months prior to Screening
* Female subjects who are not postmenopausal for at least 1 year, surgically sterile (does not include tubal ligation), or willing to practice effective contraception (as defined by the Investigator) during the study
* Women who are breastfeeding, pregnant, or planning to become pregnant while on study
* Current enrollment in any other study treatment or disease study
* Unwillingness or inability to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the study protocol
* Subjects with walking impairment due to causes other than MS
* Other unspecified reasons that, in the opinion of the Investigator and/or Biogen Idec, make the subject unsuitable for enrollment into this study

NOTE: Other eligibility criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2009-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (15):
- Biogen Idec Investigative Site, Liège, Belgium
- Biogen Idec Investigative Site, Puebla City, Mexico
- Poland (5):
  - Biogen Idec Investigative Site, Bialystok
  - Biogen Idec Investigative Site, Bydgoszcz
  - Biogen Idec Investigative Site, Lodz
  - Biogen Idec Investigative Site, Poznan
  - Biogen Idec Investigative Site, Warsaw
- Romania (2):
  - Biogen Idec Investigative Site, Bucharest
  - Biogen Idec Investigative Site, Mures
- Biogen Idec Investigative Site, Riyadh, Saudi Arabia
- Ukraine (5):
  - Biogen Idec Investigative Site, Dnipropetrovsk
  - Biogen Idec Investigative Site, Kharkiv
  - Biogen Idec Investigative Site, Kyiv
  - Biogen Idec Investigative Site, Lviv
  - Biogen Idec Investigative Site, Simferopol

REFERENCES:
- [Background] Voloshyna N, Havrdova E, Hutchinson M, Nehrych T, You X, Belachew S, Hotermans C, Paes D. Natalizumab improves ambulation in relapsing-remitting multiple sclerosis: results from the prospective TIMER study and a retrospective analysis of AFFIRM. Eur J Neurol. 2015 Mar;22(3):570-7. doi: 10.1111/ene.12618. Epub 2014 Dec 15. PMID 25511792

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Natalizumab
Started | 224 (number enrolled)
Safety Analysis Population | 218 (participants who had ≥1 infusion of natalizumab during the study)
Efficacy Analysis Population | 215 (participants who had ≥1 infusion of natalizumab and completed at least 1 on-treatment evaluation)
Completed | 197
Not Completed | 27
Not completed — Enrolled But Not Treated | 6
Not completed — Withdrawal by Subject | 9
Not completed — Adverse Event | 6
Not completed — Voluntary Discontinuation | 4
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Efficacy Analysis Population (participants who had at least 1 infusion of natalizumab and completed at least 1 on-treatment evaluation)
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 78

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Timed 100-meter Walk Test (T100T)
Description: In the T100T, the participant is instructed to walk as fast as possible for a distance of 100 meters.
Time Frame: Baseline, Week 24, Week 48
Population: Efficacy Analysis Population (participants who had at least 1 infusion of natalizumab and completed at least 1 on-treatment evaluation); n=number of participants with data at given time point.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
seconds
  Baseline; n=215 | 86.0 [63.7 to 128.9]
  Change from Baseline at Week 24; n=207 | -1.2 [-11.6 to 1.9]
  Change from Baseline at Week 48; n=199 | -1.6 [-13.7 to 2.8]
Statistical Analysis 1: Comparison: Natalizumab; Baseline, Week 24; Test type: Superiority or Other; p = 0.0003, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Natalizumab; Baseline, Week 48; Test type: Superiority or Other; p = 0.0002, Wilcoxon signed rank test

2. Primary Outcome: Change From Baseline in the Timed 25-foot Walk Test (T25FW)
Description: In the T25FW, the participant is instructed to walk as fast as possible for a distance of 25 feet.
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
seconds
  Baseline; n=215 | 6.6 [5.2 to 10.2]
  Change from Baseline at Week 24; n=207 | -0.1 [-0.7 to 0.2]
  Change from Baseline at Week 48; n=199 | -0.1 [-0.6 to 0.3]
Statistical Analysis 1: Comparison: Natalizumab; Baseline, Week 24; Test type: Superiority or Other; p = 0.0148, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Natalizumab; Baseline, Week 48; Test type: Superiority or Other; p = 0.0119, Wilcoxon signed rank test

3. Primary Outcome: Change From Baseline in Maximum Walking Distance (MWD)
Time Frame: Baseline, Week 24, Week 48
Population: Efficacy Analysis Population (participants who had at least 1 infusion of natalizumab and completed at least 1 on-treatment evaluation); n=those participants with observed data at given time point.
Measure: Median (Inter-Quartile Range); unit: meters
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
meters
  Baseline; n=143 | 350.0 [200.0 to 1000]
  Change from Baseline at Week 24; n=136 | 0.0 [0.0 to 170.0]
  Change from Baseline at Week 48; n=129 | 0.0 [0.0 to 150.0]
Statistical Analysis 1: Comparison: Natalizumab; Baseline, Week 24; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Natalizumab; Baseline, Week 48; Test type: Superiority or Other; p = 0.0157, Wilcoxon signed rank test

4. Primary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS)
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
units on a scale
  Baseline; n=215 | 4.0 [2.5 to 5.0]
  Change from Baseline at Week 24; n=207 | 0.0 [-0.5 to 0.0]
  Change from Baseline at Week 48; n=199 | 0.0 [-0.5 to 0.0]
Statistical Analysis 1: Comparison: Natalizumab; Baseline, Week 24; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test
Statistical Analysis 2: Comparison: Natalizumab; Baseline, Week 48; Test type: Superiority or Other; p < 0.0001, Wilcoxon signed rank test

5. Secondary Outcome: Correlation Between the EDSS and MWD (Pearson Correlation Coefficient)
Description: Pearson correlation coefficient is a measure of the linear correlation (dependence) between 2 variables, giving a value between +1 and -1 inclusive, where 1 is total positive correlation, 0 is no correlation, and -1 is total negative correlation.
Time Frame: Baseline, Week 24, Week 48
Population: Efficacy Analysis Population (participants who had at least 1 infusion of natalizumab and completed at least 1 on-treatment evaluation); n=number of participants with data evaluated at given time point.
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=143 | -0.7245
  Change from Baseline at Week 24; n=131 | -0.6937
  Change from Baseline at week 48; n=124 | -0.4188
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Pearson Correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Pearson Correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Pearson Correlation

6. Secondary Outcome: Correlation Between the EDSS and MWD (Spearman Correlation Coefficient)
Description: Spearman correlation coefficient is a non-parametric measure of the correlation (dependence) between 2 variables, giving a value between +1 and -1 inclusive, where 1 is total positive correlation, 0 is no correlation, and -1 is total negative correlation.
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 5
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=143 | -0.9197
  Change from Baseline at Week 24; n=131 | -0.6797
  Change from Baseline at week 48; n=124 | -0.5861
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Spearman correlation

7. Secondary Outcome: Correlation Between the T100T and T25FW (Pearson Correlation Coefficient)
Description: as for outcome 5
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 5
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=215 | 0.9235
  Change from Baseline at Week 24; n=207 | 0.4752
  Change from Baseline at week 48; n=199 | 0.4827
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Pearson Correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Pearson Correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Pearson Correlation

8. Secondary Outcome: Correlation Between the T100T and T25FW (Spearman Correlation Coefficient)
Description: as for outcome 6
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 5
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=215 | 0.8737
  Change from Baseline at Week 24; n=207 | 0.5558
  Change from Baseline at Week 48; n=199 | 0.4777
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Spearman correlation

9. Secondary Outcome: Correlation Between the EDSS and T25FW (Pearson Correlation Coefficient)
Description: as for outcome 5
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 5
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=215 | 0.5134
  Change from Baseline at Week 24; n=207 | 0.1945
  Change from Baseline at Week 48; n=199 | 0.1237
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Pearson Correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Pearson Correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Pearson Correlation

10. Secondary Outcome: Correlation Between the EDSS and T25FW (Spearman Correlation Coefficient)
Description: as for outcome 6
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 5
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=215 | 0.7574
  Change from Baseline at Week 24; n=207 | 0.2623
  Change from Baseline at Week 48; n=199 | 0.2661
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Spearman correlation

11. Secondary Outcome: Correlation Between the EDSS and T100T (Pearson Correlation Coefficient)
Description: as for outcome 5
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 5
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=215 | 0.5356
  Change from Baseline at Week 24; n=207 | 0.2176
  Change from Baseline at Week 48; n=199 | 0.1218
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Pearson Correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p = 0.0016, Pearson Correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p = 0.0866, Pearson Correlation

12. Secondary Outcome: Correlation Between the EDSS and T100T (Spearman Correlation Coefficient)
Description: as for outcome 6
Time Frame: Baseline, Week 24, Week 48
Population: as for outcome 5
Measure: Number; unit: Correlation coefficient
Arm/Group | Natalizumab
Number analyzed (Participants) | 215
Correlation coefficient
  Baseline; n=215 | 0.7269
  Change from Baseline at Week 24; n=207 | 0.3778
  Change from Baseline at Week 48; n=199 | 0.2898
Statistical Analysis 1: Comparison: Natalizumab; Baseline; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 2: Comparison: Natalizumab; Change from Baseline at Week 24; Test type: Superiority or Other; p < 0.0001, Spearman correlation
Statistical Analysis 3: Comparison: Natalizumab; Change from Baseline at Week 48; Test type: Superiority or Other; p < 0.0001, Spearman correlation

13. Secondary Outcome: Improvement in Timed 25FT Walk Speed and T100T Speed at Week 24 and 48
Description: To determine how well each of the walking tests, T100T or T25FW, predicts walking limitations, participants were stratified by baseline EDSS scores, and walking tests at Weeks 24 and 48 were analyzed. A 15% or 20% improvement indicates that, when compared with baseline walking speed (meters per second), there is at least 15% or 20% improvement at the corresponding timepoint, e.g. (speed at Week 24 - speed at baseline)/speed at baseline*100% ≥ 15% or 20%. Confirmed (conf) improvement at Week 48 indicates that the participant has at least 15% (or 20%) improvement in walking speed at both Week 24 and Week 48.
Time Frame: Baseline, Week 24, Week 48
Population: Efficacy Analysis Population (participants who had at least 1 infusion of natalizumab and completed at least 1 on-treatment evaluation); n= number of participants with evaluable data at time point.
Measure: Number; unit: participants
Groups:
- Natalizumab: Baseline EDSS 0 to 2.5: natalizumab 300 mg IV every 4 weeks for 48 weeks in participants with a Baseline EDSS of 0 to 2.5
- Natalizumab: Baseline EDSS 3.0 to 4.0: natalizumab 300 mg IV every 4 weeks for 48 weeks in participants with a Baseline EDSS 3.0 to 4.0
- Natalizumab: Baseline EDSS >= 4.5: natalizumab 300 mg IV every 4 weeks for 48 weeks in participants with a Baseline EDSS >= 4.5
Arm/Group | Natalizumab: Baseline EDSS 0 to 2.5 | Natalizumab: Baseline EDSS 3.0 to 4.0 | Natalizumab: Baseline EDSS >= 4.5
Number analyzed (Participants) | 53 | 74 | 80
participants
  T25FW: 15% Improved at Week 24; n=53,74,80 | 6 | 11 | 19
  T25FW: 15% Improved at Week 48; n=52,74,73 | 8 | 12 | 15
  T25FW: 15% Improved at Week 48 conf; n=52,74,72 | 3 | 6 | 10
  T25FW: 20% Improved at Week 24; n=52,74,80 | 5 | 8 | 14
  T25FW: 20% Improved at Week 48; n=52,74,73 | 6 | 8 | 12
  T25FW: 20% Improved at Week 48 conf; n=52,74,72 | 2 | 4 | 7
  T100T: 15% Improved at Week 24; n=53,74,80 | 11 | 13 | 24
  T100T: 15% Improved at Week 48; n=52,74,73 | 11 | 20 | 24
  T100T: 15% Improved at Week 48 conf; n=52,74,72 | 7 | 12 | 21
  T100T: 20% Improved at Week 24; n=53,74,80 | 10 | 10 | 18
  T100T: 20% Improved at Week 48; n=52,74,73 | 9 | 17 | 23
  T100T: 20% Improved at Week 48 conf; n=52,74,72 | 6 | 9 | 16

ADVERSE EVENTS:
Time Frame: Day 1 (Baseline) through Week 48 (± 7 days) plus 4 weeks (± 7 days) follow-up
Arm/Group | Natalizumab
Serious Adverse Events (participants affected / at risk) | 7/218
Other Adverse Events (participants affected / at risk) | 28/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=218)
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Sudden death (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab (N=218)
Upper respiratory tract infection (Infections and infestations) | 18
Headache (Nervous system disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.